CLINICAL TRIAL: NCT01391013
Title: A Randomised, Controlled, Open-Label Trial to Compare Brachial Artery Reactivity and Cardiovascular Risk of a Treatment Simplification by Darunavir/Ritonavir (DRV/r) 800/100 mg O.D. Versus a Triple Combination Therapy Containing DRV/r in HIV-1 Infected Subjects With Undetectable Plasma HIV-1 RNA on Their Current Treatments.
Brief Title: A Study to Compare Brachial Artery Reactivity and Cardiovascular Risk of a Treatment Simplification by Darunavir/Ritonavir (DRV/r) 800/100 mg Versus a Triple Combination Therapy Containing DRV/r in HIV-1 Infected Patients
Acronym: MONARCH
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen-Cilag S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR017575; TMC114HIV3017 (Other: Janssen-Cilag S.p.A., Italy); TMC-C-07-IT-016 (Other: Janssen-Cilag S.p.A., Italy)
Record Dates: First submitted 2011-06-23; First posted 2011-07-11 (Estimated); Results first posted 2013-06-27 (Estimated); Last update posted 2013-06-27 (Estimated); Status verified 2013-05

CONDITIONS: Human Immunodeficiency Virus 1
Keywords: Human immunodeficiency virus 1; Acquired immunodeficiency syndrome; Immunologic deficiency syndrome; Darunavir/ritonavir; Darunavir; Ritonavir; Nucleoside reverse transcriptase inhibitors (NRTIs); Prezista
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Immunologic Deficiency Syndromes | interventions — Darunavir; Ritonavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Monotherapy (Experimental): Monotherapy: darunavir/ritonavir (DRV/r) will be administered for 48 weeks.
  Interventions: Drug: Darunavir(DRV); Drug: Ritonavir
- Combination therapy (Experimental): DRV/r along with 2 nucleoside reverse transcriptase inhibitors (NRTIs) will be administered for 48 weeks and whenever possible, participants should take these medications at the same time. Switch of NRTIs will be allowed in the event of suspected toxicity/intolerance, providing this change can be linked to a documented adverse event (AE)/serious AE.
  Interventions: Drug: Darunavir(DRV); Drug: Ritonavir; Drug: 2 nucleoside reverse transcriptase inhibitors (NRTIs)

INTERVENTIONS:
Drug: Darunavir(DRV) — Oral administration of tablet DRV 800 mg (2 tablets of 400 mg) once daily at the same time, within 30 minutes after food for 48 weeks
  Other Names: Prezista
Drug: Ritonavir — Oral administration of tablet ritonavir 100 mg once daily at the same time, within 30 minutes after food for 48 weeks
Drug: 2 nucleoside reverse transcriptase inhibitors (NRTIs) — 2 NRTIs will be administered as per the package inserts.
  Arms: Combination therapy

SUMMARY:
The purpose of this study is to compare change of brachial artery flow mediated vasodilatation using Darunavir/Ritonavir (DRV/r) 800/100 mg once daily as a monotherapy (use of a single medication) versus a triple combination therapy containing 2 nucleoside reverse transcriptase inhibitors (NRTIs) and DRV/r in Human immunodeficiency virus-1 (HIV-1) infected participants.

DETAILED DESCRIPTION:
This is a Phase II, randomized (the study medication is assigned by chance), open-label (all people know the identity of the intervention), controlled, single centre study. The study consists of 3 phases including, the screening phase (4 weeks before administration of study medication), treatment phase (48 weeks), and the follow-up phase (4 weeks). In the treatment phase, HIV-infected participants who have not changed their first-line treatment of highly active antiretroviral therapy (HAART) for at least 8 weeks and have documented evidence of their HIV- ribonucleic acid (RNA) measurements being virologically suppressed (HIV-RNA less than 50 copies/mL) for at least 24 weeks prior to the screening, will be randomly assigned equally in two treatment arms: triple combination therapy arm (DRV/r 800/100 mg once daily plus 2 NRTIs) or monotherapy arm (DRV/r 800/100 mg once daily). Participants in the triple combination arm who are already on 2 NRTIs prior to randomization may remain on these or switch them at baseline, where the participants on the monotherapy arm will discontinue HAART at baseline and will start DRV/r 800/100 mg once daily. Safety evaluations will include assessment of adverse events, significant vital signs, and significant laboratory tests. The total duration of the study will be 56 weeks.

ELIGIBILITY:
Inclusion Criteria: - Human immunodeficiency virus-1 (HIV-1) infected participants on their first-line treatment with highly active antiretroviral therapy (HAART) (combination of 2 or 3 nucleoside reverse transcriptase inhibitors [NRTIs] with at least 1 additional antiretroviral [ARV] from the non-nucleoside reverse transcriptase inhibitor [NNRTI] and/or protease inhibitors [PI] class) for at least 24 weeks, provided the same ARV combination for at least 8 weeks before screening

* Participants' preference for a more convenient regimen and/or any current or history of toxicity on actual regimen
* Plasma HIV-1 ribonucleic acid (RNA) less than 50 cp/ml for at least 24 weeks before screening, where single viral blips of more than 50 copies/mL are allowed
* Cluster of differentiation 4 (CD4) count more than 100/mm3 at the start of HAART and more than 200/mm3 at screening
* Healthy on the basis of physical examination, medical history, vital signs, clinical laboratory tests, and 12-lead electrocardiogram performed at screening
* Agrees to protocol-defined use of effective contraception
* Postmenopausal, surgically sterile, or abstinent female participants

Exclusion Criteria:

* History of coronary heart disease, uncontrolled hypertension, peripheral vascular disease and or cerebrovascular disease
* History of virological failure on highly active antiretroviral therapy, plasma HIV-1 ribonucleic acid more than 500 copies/mL after initial full virological suppression while on ARV therapy and any PI mutations
* Participants with significantly hepatic and liver insufficiency or diagnosed with acute viral hepatitis or have active clinically significant diseases and acquired immune deficiency syndrome (AIDS) defining illness at screening
* Current significant tobacco use, active drug or alcohol use or dependence
* Use of lipid-lowering drugs within 4 weeks prior to study entry and use of testosterone, anabolic steroids, oral contraceptives or hormonal replacement within 12 weeks prior to study entry or previous or current use of darunavir
* Use of systemic glucocorticoids, long-acting inhaled steroids (inhaled via mouth or nose), or other immunomodulators within 30 days prior to study entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2009-06; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag S.p.A. Clinical Trial, Study Director — Janssen-Cilag S.p.A.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 30 participants were enrolled at a single site in Italy.
Pre-assignment Details: 30 participants were randomly assigned to 2 treatment groups (15 participants in each group) and all participants received the study medication.
Groups:
- Monotherapy: 2 tablets of darunavir (2 X 400 mg) and 1 tablet ritonavir (100 mg) administered once daily
- Combination Therapy: 2 tablets of darunavir (2 X 400 mg) and 1 tablet ritonavir (100 mg) once daily + 2 nucleoside reverse transcriptase inhibitors (NRTIs)
Period: Overall Study
Arm/Group | Monotherapy | Combination Therapy
Started | 15 | 15
Completed | 15 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Monotherapy | Combination Therapy | Total
Number analyzed (Participants) | 15 | 15 | 30
Age Continuous [Median (Inter-Quartile Range); unit: Years] | 44.8 [34.5 to 55.1] | 43.0 [35.0 to 46.8] | 44.6 [35.0 to 47.4]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 7
  Male | 12 | 11 | 23
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 14 | 15 | 29
  Black | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 24 in Brachial Artery Flow Mediated Vasodilatation (FMD): Median Change in FMD (%)
Description: Brachial artery FMD is calculated as the percentage increase in brachial artery diameter with hyperemia (an increase in the quantity of blood flow to a body part) induced relative to the resting brachial artery diameter. Percentage of brachial artery diameter is measured as FMD diameter/basal diameter.
Time Frame: Baseline (Day 1 of Week 1) to Week 24
Population: Participants who were randomized, who received the study medication, and who contributed any efficacy data after the start of study treatment.
Measure: Median (Inter-Quartile Range); unit: Percentage of brachial artery diameter
Arm/Group | Monotherapy | Combination Therapy
Number analyzed (Participants) | 15 | 15
Percentage of brachial artery diameter | -4.8 [-7.0 to 0.3] | -0.6 [-4.7 to 3.3]
Statistical Analysis 1: Comparison: Monotherapy vs Combination Therapy; Test type: Superiority or Other; p = 0.08, Nonparametric Wilcoxon rank sum test

2. Secondary Outcome: Change From Baseline to Week 48 in Brachial Artery FMD: Median Change in FMD (%)
Description: Brachial artery FMD is calculated as the percentage increase in brachial artery diameter with hyperemia induced relative to the resting brachial artery diameter. Percentage of brachial artery diameter is measured as FMD diameter/basal diameter.
Time Frame: Baseline to Week 48
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Percentage of brachial artery diameter
Arm/Group | Monotherapy | Combination Therapy
Number analyzed (Participants) | 15 | 15
Percentage of brachial artery diameter | -4.4 [-6.2 to 2.6] | -3 [-4.5 to 4.0]
Statistical Analysis 1: Comparison: Monotherapy vs Combination Therapy; Test type: Superiority or Other; p = 0.88, Nonparametric Wilcoxon rank sum test

3. Secondary Outcome: Number of Participants With a Human Immunodeficiency Virus- Ribonucleic Acid (HIV-RNA) Greater Than or Equal to 50 Copies/mL
Time Frame: Screening (Week -4), Week 1 (Day 1), Week 4, Week 12, Week 24, Week 36, Week 48, and follow-up (Week 52)
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Monotherapy | Combination Therapy
Number analyzed (Participants) | 15 | 15
Participants
  Screening (Week -4) | 0 [-6.2 to 2.6] | 0 [-4.5 to 4.0]
  Week 1 (Day 1) | 1 | 0
  Week 4 | 0 | 0
  Week 12 | 0 | 1
  Week 24 | 0 | 1
  Week 36 | 2 | 0
  Week 48 | 1 | 0
  Follow up (Week 52) | 2 | 0
Statistical Analysis 1: Comparison: Monotherapy vs Combination Therapy; Test type: Superiority or Other; p = 0.31, Nonparametric Wilcoxon rank sum test; This statistical analysis applies to 'Week 48'

4. Secondary Outcome: Change From Baseline to Week 48 in Circulating Endothelial Cells
Time Frame: Baseline to Week 48
Population: as for outcome 1
Measure: Median (Full Range); unit: Endothelial cells
Arm/Group | Monotherapy | Combination Therapy
Number analyzed (Participants) | 15 | 15
Endothelial cells
  Baseline | 5.09 [0 to 105.6] | 14.6 [0 to 551.4]
  Week 48 | 37 [0 to 5533] | 64 [0 to 4256]
Statistical Analysis 1: Comparison: Monotherapy vs Combination Therapy; Test type: Superiority or Other; p = 0.37, Nonparametric Wilcoxon rank sum test; This statistical analysis applies to 'Week 48'

5. Secondary Outcome: Change From Baseline to Week 48 in Precursors of Circulating Endothelial Cells
Time Frame: Baseline to Week 48
Population: as for outcome 1
Measure: Median (Full Range); unit: Endothelial cells
Arm/Group | Monotherapy | Combination Therapy
Number analyzed (Participants) | 15 | 15
Endothelial cells
  Baseline | 16 [0 to 60] | 18 [0 to 93]
  Week 48 | 120 [0 to 519] | 108 [0 to 715]
Statistical Analysis 1: Comparison: Monotherapy vs Combination Therapy; Test type: Superiority or Other; p = 0.66, Nonparametric Wilcoxon rank sum test; This statistical analysis applies to 'Week 48'

6. Secondary Outcome: Change From Baseline in Mean Low-density Lipoprotein (LDL) Cholesterol at Week 24 and Week 48: Median Change in LDL
Time Frame: Baseline (Day1 of Week 1), Week 24, and Week 48
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Monotherapy | Combination Therapy
Number analyzed (Participants) | 15 | 15
mg/dL
  Week 24 | 17 [0 to 40] | 6 [-17 to 20]
  Week 48 | 14 [7 to 42] | 5 [-12 to 19]
Statistical Analysis 1: Comparison: Monotherapy vs Combination Therapy; Test type: Superiority or Other; p = 0.02, Nonparametric Wilcoxon rank sum test; This statistical analysis applies to 'Week 48'

7. Secondary Outcome: Change From Baseline in Mean High-density Lipoprotein (HDL) Cholesterol at Week 24 and Week 48: Median Change in HDL
Time Frame: Baseline, Week 24, and Week 48
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Monotherapy | Combination Therapy
Number analyzed (Participants) | 15 | 15
mg/dL
  Week 24 | -1 [-6 to 3] | -6 [-9 to 4]
  Week 48 | -4 [-5 to 0] | -6 [-11 to -1]
Statistical Analysis 1: Comparison: Monotherapy vs Combination Therapy; Test type: Superiority or Other; p = 0.12, Nonparametric Wilcoxon rank sum test; This statistical analysis applies to 'Week 48'

8. Secondary Outcome: Change From Baseline in Mean Triglycerides at Week 24 and Week 48: Median Change in Triglycerides
Time Frame: Baseline, Week 24, and Week 48
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Monotherapy | Combination Therapy
Number analyzed (Participants) | 15 | 15
mg/dL
  Week 24 | 15 [-18 to 42] | -1 [-28 to 25]
  Week 48 | 24 [-15 to 64] | 6 [-8 to 38]
Statistical Analysis 1: Comparison: Monotherapy vs Combination Therapy; Test type: Superiority or Other; p = 0.71, Nonparametric Wilcoxon rank sum test; This statistical analysis applies to 'Week 48'

9. Secondary Outcome: Change From Baseline in Insulin Sensitivity at Week 24 and Week 48: Median Change in Homeostasis Model Assessment of Insulin Resistance (HOMA-IR)
Description: The Homeostatic Model Assessment (HOMA) is a method used to quantify insulin resistance and beta-cell function. HOMA-IR is reflected in the diminished effect of insulin on hepatic glucose production. HOMA-IR is calculated as: (Glucose [mg/dL] X Insulin [pmol/L]) / (405 X 6.945). Higher scores indicate worse insulin resistance.
Time Frame: Baseline, Week 24, and Week 48
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: HOMA score
Arm/Group | Monotherapy | Combination Therapy
Number analyzed (Participants) | 15 | 15
HOMA score
  Week 24 | -0.2 [-1.4 to 0.6] | -0.3 [-1.1 to 0.3]
  Week 48 | -0.6 [-1.1 to 0.0] | -0.5 [-1.6 to -0.1]
Statistical Analysis 1: Comparison: Monotherapy vs Combination Therapy; Test type: Superiority or Other; p = 0.83, Nonparametric Wilcoxon rank sum test; This statistical analysis applies to 'Week 48'

10. Secondary Outcome: Change From Baseline in Mean Framingham Risk Score at Week 24 and Week 48: Medican Change in Framingham Risk Score
Description: The Framingham Risk Score is used to estimate the 10-year cardiovascular risk of a participant. It is calculated according to age, laboratory values of total cholesterol and HDL cholesterol, smoking status, and systolic blood pressure. The framingham risk score is calculated as: for males: 0 point (1 percentage) up to 17 points (30 percentages); whereas for females: 0 to 9 points (1 percentage) up to 25 points (30 percentage). Higher scores indicate high cardiovascular risk.
Time Frame: Baseline, Week 24, and Week 48
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Framingham risk score
Arm/Group | Monotherapy | Combination Therapy
Number analyzed (Participants) | 15 | 15
Framingham risk score
  Week 24 | 0 [0 to 1] | 0 [-1 to 3]
  Week 48 | 1 [0 to 2] | 1 [0 to 3]
Statistical Analysis 1: Comparison: Monotherapy vs Combination Therapy; Test type: Superiority or Other; p = 0.66, Nonparametric Wilcoxon rank sum test; This statistical analysis applies to 'Week 48'

11. Secondary Outcome: Change From Baseline to Week 48 in Leg Fat Content: Median Change in Leg Fat (Total)
Description: Leg fat content will be analyzed by Dual Energy X-ray Absortiometry (DEXA scan).
Time Frame: Baseline to Week 48
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Percentage of fat
Arm/Group | Monotherapy | Combination Therapy
Number analyzed (Participants) | 15 | 15
Percentage of fat | -57 [-447 to 419] | -288 [-794 to 601]
Statistical Analysis 1: Comparison: Monotherapy vs Combination Therapy; Test type: Superiority or Other; p = 0.76, Nonparametric Wilcoxon rank sum test

12. Secondary Outcome: Change From Baseline to Week 48 in Visceral Fat Content in Abdomen: Median Change in Visceral Abdominal Tissue (VAT)
Description: Visceral fat content in abdomen will be analyzed with median change in VAT by an abdomen Computerized Tomography.
Time Frame: Baseline to Week 48
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: cm square
Arm/Group | Monotherapy | Combination Therapy
Number analyzed (Participants) | 15 | 15
cm square | -4 [-38 to 4] | -4 [-15 to 19]
Statistical Analysis 1: Comparison: Monotherapy vs Combination Therapy; Test type: Superiority or Other; p = 0.56, Nonparametric Wilcoxon rank sum test

13. Secondary Outcome: Change From Baseline to Week 48 in Femoral Neck T Score: Median Change in Femoral Neck T Score
Description: T score is used to calculate bone mineral density (calcium and other types of minerals) in an area of the bone. T score is the number of standard deviations above or below the mean for a healthy 30 year old adult of the same sex and ethnicity as a participant. This score is calculated from participant's age, gender and race and skeletal site. T score has a mean of '50' and a standard deviation of '10'. T score lower than its mean indicate low bone mineral density.
Time Frame: Baseline to Week 48
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: T score
Arm/Group | Monotherapy | Combination Therapy
Number analyzed (Participants) | 15 | 15
T score | 0.2 [-0.1 to 0.4] | -0.1 [-0.2 to 0.2]
Statistical Analysis 1: Comparison: Monotherapy vs Combination Therapy; Test type: Superiority or Other; p = 0.11, Nonparametric Wilcoxon rank sum test

14. Secondary Outcome: Change From Baseline to Week 48 in Femoral Neck Z Score: Median Change in Femoral Neck Z Score
Description: Z score is used to calculate bone mineral density (calcium and other types of minerals) in an area of the bone. Z score is the number of standard deviations above or below the mean for the participant's age, sex and ethnicity. This score is calculated from participant's age, gender and race and skeletal site. Z score has a mean of '0' and a standard deviation of '1'. Z score lower than its mean indicate low bone mineral density.
Time Frame: Baseline to Week 48
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Z score
Arm/Group | Monotherapy | Combination Therapy
Number analyzed (Participants) | 15 | 15
Z score | 0.2 [-0.1 to 0.4] | 0.0 [-0.1 to 0.2]
Statistical Analysis 1: Comparison: Monotherapy vs Combination Therapy; Test type: Superiority or Other; p = 0.18, Nonparametric Wilcoxon rank sum test

15. Secondary Outcome: Change From Baseline to Week 48 in Lumbar T Score: Median Change in Lumbar T Score
Description: as for outcome 13
Time Frame: Baseline to Week 48
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: T score
Arm/Group | Monotherapy | Combination Therapy
Number analyzed (Participants) | 15 | 15
T score | 0.1 [0.0 to 0.3] | 0.0 [-0.2 to 0.1]
Statistical Analysis 1: Comparison: Monotherapy vs Combination Therapy; Test type: Superiority or Other; p = 0.03, Nonparametric Wilcoxon rank sum test

16. Secondary Outcome: Change From Baseline to Week 48 in Lumbar Z Score: Median Change in Lumbar Z Score
Description: as for outcome 14
Time Frame: Baseline to Week 48
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Z score
Arm/Group | Monotherapy | Combination Therapy
Number analyzed (Participants) | 15 | 15
Z score | 0.1 [0.0 to 0.3] | 0.0 [-0.2 to 0.1]
Statistical Analysis 1: Comparison: Monotherapy vs Combination Therapy; Test type: Superiority or Other; p = 0.04, Nonparametric Wilcoxon rank sum test

17. Secondary Outcome: Change From Baseline in Cluster of Differentiation 4 (CD4) Count Over Week 48
Time Frame: Screening (Week -4), Week 1 (Day 1), Week 4, Week 12, Week 24, Week 36, Week 48, and follow-up (Week 52)
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: CD4 cells
Arm/Group | Monotherapy | Combination Therapy
Number analyzed (Participants) | 15 | 15
CD4 cells
  Week 24 | 6 [-48 to 58] | -12 [-67 to 70]
  Week 48 | 100.1 [32 to 135] | 60 [-69 to 122]

ADVERSE EVENTS:
Time Frame: 52 weeks
Arm/Group | Monotherapy | Combination Therapy
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 10/15 | 11/15
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Monotherapy (N=15) | Combination Therapy (N=15)
Diarrhoea (Gastrointestinal disorders) | 1 | 3
Malaise (General disorders) | 1 | 1
Pyrexia (General disorders) | 3 | 1
Influenza (Infections and infestations) | 2 | 1
Blood cholesterol increased (Investigations) | 4 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 2
Blood triglycerides increased (Investigations) | 1 | 1
Low density lipoprotein increased (Investigations) | 4 | 0
Headache (Nervous system disorders) | 1 | 1
Insomnia (Psychiatric disorders) | 2 | 0
Hypertension (Vascular disorders) | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days